CLINICAL TRIAL: NCT01563809
Title: The Relationship Between Basal Androgen Levels and the Needing of LH for Controlled Ovarian Stimulation for in Vitro Fertilization
Brief Title: Basal Androgens and LH Needing for Ovarian Stimulation for in Vitro Fertilization
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Principal Investigator, Ernesto Bosch, Medical Director IVI Valencia, Instituto Valenciano de Infertilidad, IVI VALENCIA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0711-E-39-EB
Record Dates: First submitted 2012-03-22; First posted 2012-03-27 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low androgens FSH+LH (Active Comparator): Patients with androgens below threshold receiving FSH+LH for ovarian stimulation
  Interventions: Drug: FSH+LH
- High androgens FSH+LH (Active Comparator): Patients with androgens above threshold receiving FSH+LH for ovarian stimulation
  Interventions: Drug: FSH+LH
- High androgens FSH alone (No Intervention)
- Low androgens, FSH alone (No Intervention)

INTERVENTIONS:
Drug: FSH+LH — 75 IU of LH will be given from stimulation day 1
  Arms: Low androgens FSH+LH
Drug: FSH+LH — 75 IU of LH will be given from stimulation day 1
  Arms: High androgens FSH+LH

SUMMARY:
Basing the investigators study on the evidence that basal serum androgens decrease with age, the investigators hypothesize that women with serum androgens below a certain level could be the population obtaining a benefit of Luteinizing Hormone (LH) supplementation. The objective of the present study is to explore the relationship between basal serum androgen levels and the need of LH for Controlled Ovarian Stimulation (COS) in IVF.

DETAILED DESCRIPTION:
Design: Single centre, open label, randomized controlled trial.

* Population: Patients with indication of In Vitro Fertilization (IVF) with the following criteria:
* Protocol: All patients are tested on day 3-5 of cycle for total Testosterone (Te), Dehydroepiandrosetnodione sulphate (DHEAS) and Androstenodione (Δ4). Samples are frozen and stored at -20ºC for later analysis. FSH, LH, E2, PRL and TSH are also determined. All patients follow Controlled Ovarian Stimulation for IVF with a GnRH agonist long protocol. They are randomized to receive recombinant (r) FSH alone (225 IU/day) or r-FSH + r-LH (225+75 IU/day).
* Sample size calculation: To detect a difference from 40 to 60% (Relative risk: 1.50) on pregnancy rate (PR) between patients with low and high androgen levels with respect to the mean of each COS protocol, with a confidence level of 95% (error α=0.05) and 80% of power (error β=0.2), 97 patients per arm were needed. (n=388 patients). Rounding up, 400 patients are to be recruited.

ELIGIBILITY:
Inclusion Criteria:

* 1st-2nd IVF cycle
* Regular cycle (25-35 days)
* Age 18 - 42
* BMI: 18-29.9

Exclusion Criteria:

* LH:FSH > 2
* Low response background (< 5 oocytes)
* Recurrent pregnancy loss
* Preimplantational genetic diagnosis indication
* Any systemic, metabolic or endocrinological disorder.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2008-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Clinical Pregnancy Rate | 45 days
  Use of rec LH supplementation for controlled ovarian stimulation for IVF

CONTACTS AND LOCATIONS:
Locations (1):
- IVI Valencia, Valencia, Spain